CLINICAL TRIAL: NCT07310485
Title: Examining the Impact of Phytoestrogens Supplementation and on the Gene Expression of Anti-Müllerian Hormone, Its Receptor, and Premenstrual Syndrome in Primenopausal Women Aged 40-55 in Jordan
Brief Title: Examining the Impact of Phytoestrogens Supplementation on the Gene Expression, and Premenstrual Syndrome in Primenopausal Women
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Hadeel Ali Ghazzawi, prof, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 353/2025; 2025-150/2024 (Other Grant/Funding Number: the university of Jordan); 32152/4/1/3 (Other: Jordanian food and drug administration)
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Apparently Healthy and Not Receiving Hormonal Therapy
Keywords: phytoestrogen, flaxseed, SDG lignans, perimenopause, PMS, gene expression
MeSH Terms: interventions — Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): Microcrystalline cellulose (Placebo), taken orally once daily for 12 weeks. The capsule is matched in size, color, and taste to the active phytoestrogen supplement.
  Interventions: Dietary Supplement: Placebo
- Intevention SDG lignans (Experimental): Dietary Supplement: SDG lignans phytoestrogen 100 mg SDG (Active Ingredient), taken orally once daily for 12 weeks
  Interventions: Dietary Supplement: SDG lignans

INTERVENTIONS:
Dietary Supplement: SDG lignans — SDG lignans phytoestrogen 100 mg SDG (Active Ingredient), taken orally once daily for 12 weeks
  Other Names: flax seed extract
  Arms: Intevention SDG lignans
Dietary Supplement: Placebo — Microcrystalline cellulose (Placebo), taken orally once daily for 12 weeks. The capsule is matched in size, color, and taste to the active SDG supplement.
  Arms: placebo

SUMMARY:
This randomized, double-blind, placebo-controlled clinical trial aims to investigate the effect of flaxseed-derived phytoestrogen supplementation on gene expression of Anti-Müllerian Hormone (AMH) and its receptor (AMHR2), as well as the experience and severity of premenstrual syndrome (PMS), among perimenopausal women aged 40-55 years in Jordan. Participants will receive either flaxseed phytoestrogen extract (secoisolariciresinol diglucoside, SDG) or placebo for 12 weeks. Changes in gene expression and PMS severity will be assessed at baseline and post-intervention to explore the potential role of phytoestrogens in modulating ovarian aging and menstrual-related symptoms.

DETAILED DESCRIPTION:
Menopause is a natural biological transition characterized by progressive ovarian aging, hormonal fluctuations, and changes in menstrual patterns. Anti-Müllerian Hormone (AMH) and its receptor (AMHR2) play central roles in ovarian folliculogenesis and are considered reliable biomarkers of ovarian reserve and reproductive aging. Reduced AMH levels have been associated with earlier onset of menopause.

Phytoestrogens are plant-derived compounds structurally similar to endogenous estrogens and are capable of interacting with estrogen receptors, exerting weak estrogenic or anti-estrogenic effects depending on the hormonal milieu. Flaxseed is one of the richest dietary sources of lignans, particularly secoisolariciresinol diglucoside (SDG), which is metabolized into bioactive enterolignans.

This study is designed as a randomized, double-blind, placebo-controlled trial to evaluate the effect of daily SDG supplementation on AMH and AMHR2 gene expression and on the experience and severity of premenstrual syndrome in perimenopausal women aged 40-55 years. Participants will be randomly assigned to receive either SDG capsules (100 mg/day) or placebo for 12 weeks. Gene expression will be assessed using salivary samples collected at baseline and post-intervention. PMS severity will be evaluated using a validated Premenstrual Syndrome Scale.

Findings from this trial may contribute to understanding the role of dietary phytoestrogens in modulating reproductive aging and menstrual-related symptoms and may support future development of personalized nutritional strategies for women approaching menopause.

ELIGIBILITY:
Inclusion Criteria:

Women aged 40-55 years Jordanian nationality Body mass index (BMI) between 19 and 29.9 kg/m² Apparently healthy and not receiving hormonal therapy -

Exclusion Criteria:

Pregnancy or lactation Use of hormonal replacement therapy or hormonal contraceptives Diagnosis of chronic metabolic, cardiovascular, liver, kidney, autoimmune, or malignant disease History of gynecological disorders or surgeries Use of dietary supplements or special diets within the previous 3 months Habitual consumption of flaxseed or phytoestrogen supplements Active bowel disease or malabsorption syndrome

-

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-01-02 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Change in Gene Expression | Time Frame: Baseline (Week 0) and End of Intervention (Week 12)

SECONDARY OUTCOMES:
change of PMS severity scale | Time Frame: Baseline (Week 0) and End of Intervention (Week 12)

CONTACTS AND LOCATIONS:
Locations (1):
- the university of Jordan, Amman, Amman Governorate, Jordan

IPD SHARING:
Plan to Share IPD: No